CLINICAL TRIAL: NCT00994370
Title: Measurement of Pro-angiogenic Markers in Patients With Hepatic Metastases Undergoing Selective Internal Radiation Therapy (SIRT)
Brief Title: Measurement of Pro-angiogenic Markers in Patients With Hepatic Metastases Undergoing SIRT
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 0220080303
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Liver Cancer
Keywords: Pro-angiogenic markers; SIRT; hepatic metastases
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be obtained at intervals based on standard of care blood draws. Each sample will be analysed for circulating indicators of angiogenesis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver cancer: Patients referred for SIRT will be considered for this investigation. These patients will predominantly have stage IV colorectal metastases with liver dominant metastases or hepatocellular carcinoma. A team of oncologists, interventional radiologists, radiation oncologists and oncologic surgeons will determine that the patients are not candidates for surgical resection or ablative therapy. The patients will then be screened to confirm the patient's eligibility to receive standard of care SIRT treatment. SIRT treatment and imaging studies included in this investigation are standard of care for the patients' liver dominant disease.

SUMMARY:
This study is being done to investigate the influence of giving radiation to the liver on tumors involving the liver. Investigator is specifically looking at this effect on the blood vessels within the tumor. This effect will be measured by studying substances in the blood that the tumors produce and that cause blood vessels to grow. The effects seen on these substances may help design other treatments to improve the results of the radiation used to treat these tumors.

DETAILED DESCRIPTION:
Subjects are invited to participate in this study that have undergone a procedure as their standard of care. This procedure is known as Selective Internal Radiation Therapy (SIRT), a procedure designed for the treatment of cancer in the liver. This includes cancer that has started in the liver as well as cancer that has spread to the liver. The purpose of the study is to collect blood samples to assess for "biological markers," or substances within the blood that may promote cancer growth by causing new blood vessels to form. This study will also use a new method of analyzing medical imaging (CT scan, PET scan) to try and better understand how cancer in the liver forms new blood vessels. SIRT is standard therapy and not part of this study. This study involves blood draws only.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-85 who have been referred for SIRT as standard of care treatment for hepatocellular carcinoma or colorectal metastases to the liver and qualify for treatment with SIRT
* Life expectancy of at least 3 months

Exclusion Criteria:

- Patients are excluded from participation in this study if they are not undergoing the SIRT procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have undergone Selective Internal Radiation Therapy for the treatment of liver cancer
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cellular and peptide pro-angiogenic markers in patients with hepatic malignancy before and after SIRT | Depending on subject's treatment schedule blood samples are drawn from Day 0 through Day 120 (120 days for whole liver treatment).
  Primary objective is to develop assays for both cellular and peptide pro-angiogenic markers and determine variability of these makers in patients with hepatic malignancy before and after Selective Internal Radiation Therapy (SIRT).

SECONDARY OUTCOMES:
Imaging based predictors | Depending on subject's treatment schedule blood samples are drawn from Day 0 through Day 120 (120 days for whole liver treatment)
  To begin to develop imaging based predictors of response to SIRT.

CONTACTS AND LOCATIONS:
Overall Officials: John L Nosher, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

REFERENCES:
- [Result] Carpizo DR, Gensure RH, Yu X, Gendel VM, Greene SJ, Moore DF, Jabbour SK, Nosher JL. Pilot study of angiogenic response to yttrium-90 radioembolization with resin microspheres. J Vasc Interv Radiol. 2014 Feb;25(2):297-306.e1. doi: 10.1016/j.jvir.2013.10.030. Epub 2013 Dec 20. PMID 24360887